CLINICAL TRIAL: NCT05548764
Title: Prevention Bundles for Surgical Site Infections (PREBUSSI): a Multi-center Observational Study.
Brief Title: Prevention Bundles for SSIs (PREBUSSI).
Status: Completed | Type: Observational
Sponsor: Maximos Frountzas (Other)
Responsible Party: Sponsor-Investigator, Maximos Frountzas, Maximos Frountzas MD MPA PhD, National and Kapodistrian University of Athens
Organization: National and Kapodistrian University of Athens (Other)
Other Study IDs: PREBUSSI 2022
Record Dates: First submitted 2022-09-17; First posted 2022-09-21 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Surgical Site Infection
Keywords: SSI; prevention; bundles; PREBUSSI
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prevention Bundles: Patients in which prevention bundles for SSIs have been implemented.
  Interventions: Procedure: Prevention Bundles for SSIs
- No Prevention Bundles: Patients in which prevention bundles for SSIs have not been implemented.

INTERVENTIONS:
Procedure: Prevention Bundles for SSIs — 10 preoperative, intraoperative and postoperative bundles that aim to decrease SSIs rate after their implementation in patients that underwent abdominal surgery.
  Groups: Prevention Bundles

SUMMARY:
Surgical site infections (SSIs) are the most complication after a surgical operation and their incidence reaches 20% worldwide. SSIs have been associated to significant morbidity and mortality, high ICU admission rates, increased length of hospital stay, high readmission rates and raised cost. However, there is no registry for SSIs in Greece so far. In addition, it has been considered that almost half of SSIs could be prevented. Therefore, several prevention strategies have been suggested by international health organizations, such as WHO and NICE, that seem to be effective. The aim of the present study is to investigate the effect of 10 prevention bundles on the rate of SSIs, as well their consequences on several financial parameters of the Greek healthcare system.

DETAILED DESCRIPTION:
* 1st phase (2 months) → SSIs rate among abdominal surgical operations and reporting of patients' demographics (gender, age, comorbidities), type of surgery (upper GI, HPB, colorectal), surgical approach (open, laparoscopic), urgency classification, operation time, cost, pathogen cultures and antibiotic sensitivity test.
* 2ο phase (10 months) → implementation of 10 prevention bundles:

  1. Antibiotic delivery 1-1.5 hours before surgical incision and repeat every 4 hours intraoperatively.
  2. Hair removal with electric hair clippers using single-use bladdes.
  3. Surgical scrub with Povidone Iodine solution 4% (Betadine Surgical Scrub)
  4. Skin preparation with chlorexidine alcohol-based antiseptic solution 2%.
  5. Intraoperative and postoperative (4-6 hours) normothermia (>36οC) using warmed forced-air blankets.
  6. Perioperative normoglycemia (Glu<200mg/dl) in diabetic patients.
  7. Single-use drapes and gowns.
  8. Surgical team glove changing by before skin incision closing.
  9. Single-layer surgical incision closure with triclosan plus antimicrobial-coated sutures.
  10. Wound irrigation (skin and subcutaneous fat) with Povidone Iodine solution (Betadine) after abdominal wall closure.
* Implementation check of 10 prevention bundles preoperatively, intraoperatively and postoperatively.
* Clinical assessment on POD 1, 3, 7 and 1 month postoperatively for SSI presence (according to WHO 2018 definition).
* Reporting of patients' demographics (gender, age, comorbidities), type of surgery (upper GI, HPB, colorectal), surgical approach (open, laparoscopic), urgency classification, operation time, length of stay, cost, pathogen cultures and antibiotic sensitivity test.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Signed consent from patient or authorized representative
3. Abdominal surgery
4. Open or laparoscopic operations

Exclusion Criteria:

1. Age < 18 years old
2. No signed consent from patient or authorized representative
3. Neck, thoracic, anal, lumbar operations
4. No closure of abdominal wall or open abdomen

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients that underwent abdominal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Incidence of SSIs | 30 days
  Rate of SSIs after implementation of prevention bundles

SECONDARY OUTCOMES:
Length of hospital stay | 30 days
  Days of hospitalization.
Cost | 30 days
  Overall cost of procedures and hospitalization.
Pathogen cultures | 30 days
  Results of pathogen cultures.
Antibiotic sensitivity test | 30 days
  Antibiotics in which cultured pathogens are sensitive.
Implementation of guidelines | 30 days
  Adoptive efficacy of the 10 preventive bundles.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos G Toutouzas, MD PhD, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- Hippocration General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shrestha B, Dunn L. The Declaration of Helsinki on Medical Research involving Human Subjects: A Review of Seventh Revision. J Nepal Health Res Counc. 2020 Jan 21;17(4):548-552. doi: 10.33314/jnhrc.v17i4.1042. PMID 32001865
- [Background] Suragul W, Rungsakulkij N, Vassanasiri W, Tangtawee P, Muangkaew P, Mingphruedhi S, Aeesoa S. Predictors of surgical site infection after pancreaticoduodenectomy. BMC Gastroenterol. 2020 Jun 26;20(1):201. doi: 10.1186/s12876-020-01350-8. PMID 32586351
- [Background] Mentor K, Ratnayake B, Akter N, Alessandri G, Sen G, French JJ, Manas DM, Hammond JS, Pandanaboyana S. Meta-Analysis and Meta-Regression of Risk Factors for Surgical Site Infections in Hepatic and Pancreatic Resection. World J Surg. 2020 Dec;44(12):4221-4230. doi: 10.1007/s00268-020-05741-6. Epub 2020 Aug 18. PMID 32812136
- [Background] Fuglestad MA, Tracey EL, Leinicke JA. Evidence-based Prevention of Surgical Site Infection. Surg Clin North Am. 2021 Dec;101(6):951-966. doi: 10.1016/j.suc.2021.05.027. PMID 34774274
- [Background] Lohsiriwat V. High Compliance With Surgical Site Infection (SSI) Prevention Bundle Reduces Incisional SSI After Colorectal Surgery. Ann Coloproctol. 2021 Jun;37(3):146-152. doi: 10.3393/ac.2020.04.10.2. Epub 2020 May 15. PMID 32674555